CLINICAL TRIAL: NCT04264481
Title: Minimally Invasive Knee Osteoarthritis Pain Control Via Adductor Canal Block Versus Intra-articular Steroid and Lignocaine Injection : a Single-blinded Controlled Trial
Brief Title: Adductor Canal Block Versus Intra-articular Steroid and Lignocaine in Knee Osteoarthritis Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Anwar Suhaimi, Senior Lecturer, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201945-7302
Record Dates: First submitted 2019-11-08; First posted 2020-02-11 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Steroids; Lidocaine

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigator blinded to intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adductor Canal Block (Experimental): Adductor Canal Block (Saphaenous Nerve Block) done under Ultrasonographic guidance with 5cc of Bupivacaine, 5cc of lidocaine diluted with 10 cc of Normal Saline
  Interventions: Procedure: Adductor Canal Block
- Intra-articular Steroid and Lignocaine (Active Comparator): Intra-articular knee joint injection of 40mg triamcinolone and 1-2cc of lidocaine
  Interventions: Procedure: Intra-Articular Steroid and Lignocaine Injection

INTERVENTIONS:
Procedure: Adductor Canal Block — Ultrasound guided perineural injection of 5cc bupivacaine, 5cc lidocaine and 10 cc Normal saline
  Other Names: Saphenous Nerve Block
  Arms: Adductor Canal Block
Procedure: Intra-Articular Steroid and Lignocaine Injection — Intra-articular injection of 40mg triamcinolone and 1-2 cc of lidocaine
  Arms: Intra-articular Steroid and Lignocaine

SUMMARY:
A prospective, single blinded interventional study will be conducted in the Rehabilitation Medicine Clinic, University Malaya Medical Center for a duration of 1 year. Eligible subjects will be enrolled from all referrals of chronic knee osteoarthritis, following computer-generated randomization they will be allocated to either Adductor Canal Block (intervention) or Intra-articular Steroid and Lignocaine (control) groups. The assessor is blinded to the intervention received, which will be performed by an experienced interventionist, not participating in randomization or data collection and analysis. Demographics of participants, duration of symptoms, Numerical Rating Score (NRS) pain score and Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire score will be recorded prior to injection, 1 week, 1 month and 3 months post injection. Mann-Whitney U tests and Chi-Square test of association will be used as appropriate to compare groups at baseline. Numerical Rating Scale (NRS) pre and post intervention will be analyzed using paired t-test. Functional outcome and Quality of Life (QoL) subset of Knee Injury and Osteoarthritis Outcome Score (KOOS) Questionnaire pre and post intervention will be analyzed using paired t-test as well

DETAILED DESCRIPTION:
BACKGROUND Knee osteoarthritis (KOA) pain is major public health issue globally causing locomotor disability affecting around 251 million people worldwide according to the Global Burden of Disease 2010 Study. In Malaysia, KOA prevalence is 10% to 20% of the elderly population and negatively affects physical function especially limitation in walking (22%), carrying objects (18.6%), and dressing (12.8%). Mild to moderate KOA pain is managed with anti-inflammatory drugs and knee replacement surgery is recommended when pharmacotherapy fails. However, 81% of the patients would refrain from undergoing surgery as it is expensive. Currently there is no effective pharmaceutical treatments for KOA pain & functional disability. Most studies with regards to adductor canal block for KOA pain are done in the immediate post-operative period with only 3 studies looking into ACB in the chronic KOA population: 1 case report and 2 retrospective studies. Thus, there is a need for head to head comparison between Adductor Canal Block (ACB) and Intra-Articular Steroid and Lignocaine (IASL).

OBJECTIVES

Primary objective:

1. Investigate the reduction in pain score following adductor canal block in comparison to intra-articular steroid and lignocaine in chronic Knee Osteoarthritis (KOA) pain.

   Secondary objectives:
2. To ascertain the functional improvement following Adductor Canal Block versus Intra-Articular Steroid and Lignocaine for chronic Knee Osteoarthritis (KOA)
3. To evaluate the Quality of life improvement following Adductor Canal Block versus Intra-Articular Steroid and Lignocaine for chronic Knee Osteoarthritis

METHOD

A prospective, single blinded interventional study will be conducted in the Rehabilitation Medicine Clinic, University Malaya Medical Center for a duration of 1 year. Eligible subjects will be enrolled from all referrals of chronic knee osteoarthritis, following computer-generated randomization they will be allocated to either Adductor Canal Block (intervention) or Intra-Articular Steroid and Lignocaine (control) groups. The assessor is blinded to the intervention received, which will be performed by an experienced interventionist, not participating in randomization or data collection and analysis. Demographics of participants, duration of symptoms, Numerical Rating Score (NRS) pain score and Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire score will be recorded prior to injection, 1 week, 1 month and 3 months post injection. Mann-Whitney U tests and Chi-Square test of association will be used as appropriate to compare groups at baseline. Numerical Rating Scale (NRS) pre and post intervention will be analyzed using paired t-test. Functional outcome and Quality of Life (QoL) subset of Knee Injury and Osteoarthritis Outcome Score (KOOS) Questionnaire pre and post intervention will be analyzed using paired t-test as well.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Knee Osteoarthritis according to criteria of American College of Rheumatology

  * Antero-medial knee pain of at least 6 months duration
  * Matching symptoms with Knee X-ray findings of KOA
  * Kellgran-Lawrence staging of 2-4
  * Pain score of at least NRS(Numerical Rating Scale) 4/10 during weight bearing

Exclusion Criteria:

* Presence of other knee diseases such as fracture or rheumatic diseases
* Referred pain from the back suggestive of lumbar radiculopathy
* Previous knee surgery
* Lateral knee pain
* History of knee joint injections (Intra-articular injections or ACB) within 3 months of study
* Neuropathic knee pain
* Unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
Knee Pain score change | Before intervention, within 1 hour, after 4 weeks, after 12 weeks (change from baseline - before intervention)
  Change from baseline Pain Score On weight Bearing using numerical rating scale (Visual Analog Scale / Numerical Rating Scale : from 0 to 10, 0 being the absence of pain with maximum score of 10 indicating most severe pain - increasing value given indicates more severe pain)

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) Questionnaire - Functional component score change | Before intervention, after 4 weeks , after 12 weeks - measuring change from baseline score (before intervention)at the intervals mentioned
  Self administered questionnaire - patients answer a series of 17 questions : answers are based on 5 responses utilizing a Likert scale and scored base on this formula 100 - [Mean Score (A1-A17)×100 / 4]
  As long as at least 50% of the subscale items are answered for each subscale, a mean score can be calculated
  The score is a percentage score from 0 to 100, with 0 representing extreme problems and 100 representing no problems
Knee Injury and Osteoarthritis Outcome Score (KOOS) Questionnaire - Quality of Life component score change | Before intervention, after 4 weeks , after 12 weeks - measuring change from baseline score (before intervention)at the intervals mentioned
  Self administered questionnaire - patients answer a series of 4 questions : answers are based on 5 responses utilizing a Likert scale and scored base on this formula 100 - [Mean Score (Q1-Q4)×100 / 4]
  As long as at least 50% of the subscale items are answered for each subscale, a mean score can be calculated
  The score is a percentage score from 0 to 100, with 0 representing extreme problems and 100 representing no problems

CONTACTS AND LOCATIONS:
Overall Officials: Anwar Suhaimi, MBBS, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Center, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neogi T. The epidemiology and impact of pain in osteoarthritis. Osteoarthritis Cartilage. 2013 Sep;21(9):1145-53. doi: 10.1016/j.joca.2013.03.018. PMID 23973124
- [Background] Vos T, Flaxman AD, Naghavi M, Lozano R, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gosselin R, Grainger R, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Ma J, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Years lived with disability (YLDs) for 1160 sequelae of 289 diseases and injuries 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2163-96. doi: 10.1016/S0140-6736(12)61729-2. PMID 23245607
- [Background] Veerapen K, Wigley RD, Valkenburg H. Musculoskeletal pain in Malaysia: a COPCORD survey. J Rheumatol. 2007 Jan;34(1):207-13. PMID 17216688
- [Background] Palazzo C, Ravaud JF, Papelard A, Ravaud P, Poiraudeau S. The burden of musculoskeletal conditions. PLoS One. 2014 Mar 4;9(3):e90633. doi: 10.1371/journal.pone.0090633. eCollection 2014. PMID 24595187
- [Background] Hochberg MC, Altman RD, April KT, Benkhalti M, Guyatt G, McGowan J, Towheed T, Welch V, Wells G, Tugwell P; American College of Rheumatology. American College of Rheumatology 2012 recommendations for the use of nonpharmacologic and pharmacologic therapies in osteoarthritis of the hand, hip, and knee. Arthritis Care Res (Hoboken). 2012 Apr;64(4):465-74. doi: 10.1002/acr.21596. PMID 22563589
- [Background] Carr AJ, Robertsson O, Graves S, Price AJ, Arden NK, Judge A, Beard DJ. Knee replacement. Lancet. 2012 Apr 7;379(9823):1331-40. doi: 10.1016/S0140-6736(11)60752-6. Epub 2012 Mar 6. PMID 22398175
- [Background] Liddle AD, Pegg EC, Pandit H. Knee replacement for osteoarthritis. Maturitas. 2013 Jun;75(2):131-6. doi: 10.1016/j.maturitas.2013.03.005. Epub 2013 Apr 9. PMID 23582106
- [Background] Koh IJ, Choi YJ, Kim MS, Koh HJ, Kang MS, In Y. Femoral Nerve Block versus Adductor Canal Block for Analgesia after Total Knee Arthroplasty. Knee Surg Relat Res. 2017 Jun 1;29(2):87-95. doi: 10.5792/ksrr.16.039. PMID 28545172
- [Background] Osteras N, van Bodegom-Vos L, Dziedzic K, Moseng T, Aas E, Andreassen O, Mdala I, Natvig B, Rotterud JH, Schjervheim UB, Vlieland TV, Hagen KB. Implementing international osteoarthritis treatment guidelines in primary health care: study protocol for the SAMBA stepped wedge cluster randomized controlled trial. Implement Sci. 2015 Dec 2;10:165. doi: 10.1186/s13012-015-0353-7. PMID 26631224
- [Background] Silva AG, Alvarelhao J, Queiros A, Rocha NP. Pain intensity is associated with self-reported disability for several domains of life in a sample of patients with musculoskeletal pain aged 50 or more. Disabil Health J. 2013 Oct;6(4):369-76. doi: 10.1016/j.dhjo.2013.04.007. Epub 2013 May 28. PMID 24060260
- [Result] Lee DH, Lee MY, Kwack KS, Yoon SH. Effect of adductor canal block on medial compartment knee pain in patients with knee osteoarthritis: Retrospective comparative study. Medicine (Baltimore). 2017 Mar;96(12):e6374. doi: 10.1097/MD.0000000000006374. PMID 28328826
- [Result] Eker HE, Cok OY, Aribogan A, Arslan G. The efficacy of intra-articular lidocaine administration in chronic knee pain due to osteoarthritis: A randomized, double-blind, controlled study. Anaesth Crit Care Pain Med. 2017 Apr;36(2):109-114. doi: 10.1016/j.accpm.2016.05.003. Epub 2016 Jul 30. PMID 27485803
- [Result] Arroll B, Goodyear-Smith F. Corticosteroid injections for osteoarthritis of the knee: meta-analysis. BMJ. 2004 Apr 10;328(7444):869. doi: 10.1136/bmj.38039.573970.7C. Epub 2004 Mar 23. PMID 15039276
- See also: 3. Ministry of Health Malaysia. Clinical Practice Guidelines on the Management of Osteoarthritis. 2010 — http://www.moh.gov.my/index.php/file_manager/dl_item/6257467262485674595851676447567961326c7561533945636d466d6446394455456466543045756347526d
- See also: Knee Pain and Functional Disability of Knee Osteoarthritis Patients Seen at Malaysian — http://www.medic.upm.edu.my/upload/dokumen/2017090710491402_MJMHS_Vol13_No2_2017_-_0016_-_p7-15_4th_proof.pdf